CLINICAL TRIAL: NCT00373568
Title: Miltefosine (42 Days) for Mucosal Leishmaniasisi
Brief Title: Miltefosine (Long Course) for Bolivian Mucosal Leishmaniasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AB Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05--01
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Leishmaniasis
Keywords: mucosal; miltefosine
MeSH Terms: conditions — Leishmaniasis | interventions — miltefosine

INTERVENTIONS:
Drug: miltefosine: 2.5 mg/kg/day for 42 days

SUMMARY:
Miltefosine (longer course) will be used to try to improve the cure rate of mucosal leishmaniasis

DETAILED DESCRIPTION:
Miltefosine (42 days) will be used to try to improve upon the cure rate with 28 days of drug for bolivian mucosal leishmaniasisi

ELIGIBILITY:
Inclusion Criteria:

* Mucosal leishmaniasis

Exclusion Criteria:

* No comcomitant disease as judged by laboratory and clinical parameters

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2005-04; Study Completion 2007-12

PRIMARY OUTCOMES:
efficacy

SECONDARY OUTCOMES:
safety

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Soto, MD, Principal Investigator — CIBIC
Locations (1):
- Palos Blancos, Palos Blancos, Bolivia